CLINICAL TRIAL: NCT05353387
Title: The Effect of the Motivational Interviewing Technique Applied to Women in the Menopause Period on Their Participation in Breast and Cervical Cancer Screenings
Brief Title: The Effect of the Motivational Interviewing Technique on Breast and Cervical Cancer Screenings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Tugba OZTURK, Principal Investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/73
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Menopause; Cervix Cancer; Breast Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group- Motivational Interviewing (Experimental): Standard protocols and participation in Motivational Interviews
  Interventions: Other: Motivational Interviewing
- Control Group (No Intervention): Standard protocols

INTERVENTIONS:
Other: Motivational Interviewing — Motivational Interviewing will be carried out in 3 different sessions, each to be conducted one week apart. 6 weeks after the last interview, first follow up would be conducted through phone communication and 6 weeks after the first follow up, a face-to-face interview would be conducted for the scales to be applied to the participants again.
  Arms: Intervention Group- Motivational Interviewing

SUMMARY:
This study will be conducted to evaluate the effect of the motivational interviewing technique applied to menopausal women on their participation in breast and cervical cancer screenings. This is a randomized controlled intervention study in which the study sample will consist of 120 menopausal women, who visit the health care centers in the city of Kutahya. There will be one intervention group with a total of 60 participants and a control group with the same number of participants. The intervention group will have motivational interviews whereas the control group participants will follow the normal protocols.

DETAILED DESCRIPTION:
This study will be conducted to evaluate the effect of the motivational interviewing technique applied to menopausal women on their participation in breast and cervical cancer screenings. This is a randomized controlled intervention study in which the study sample will consist of 120 menopausal women, who visit the health care centers in the city of Kutahya. There will be one intervention group with a total of 60 participants and a control group with the same number of participants. The intervention group will have motivational interviews whereas the control group participants will follow the normal protocols.

The Turkish version of Champion's Health Belief Model Scale and The Health Belief Model Scale for Cervical Cancer and the Pap Smear Test will be applied to all the participants in both groups.

Then for the intervention group, the motivational interviewing will be carried out in 3 different sessions, each to be conducted one week apart. 6 weeks after the last interview, first follow up would be conducted through phone communication and 6 weeks after the first follow up, a face-to-face interview would be conducted for the scales to be applied to the participants again. For the control group, the scales will be applied for the second time at the same time as the intervention group and they will be given a training manual and their questions will be answered by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Visiting any family health centers in the city of Kütahya,
* Without any cancer diagnosis and treatment,
* Not having had a clinical breast examination in the last 1 year, with no natural menstrual period in the last 1 year, have entered menopause and are 69 years old (included) maximum,
* Without a mammogram in the last 2 years in women who have gone through menopause and are 69 years old (included).
* Without an HPV or Pap smear test in the last 5 years in women who have entered menopause and are in the age range of 65 (including),
* Being literate,
* Able to communicate.

Exclusion Criteria:

* Having been diagnosed with any cancer,
* Inability to communicate,
* Failure to continue the phases of the study for any reason.

Max Age: 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Turkish Version of Champion's Health Belief Model Scale (CHBMS-T) | 4 Months Questions were answered on a 5-point Likert-type response scale ranging from 1 (strongly disagree) to 5 (strongly agree), and mean scores were computed for each subscale.
  Champion's Health Belief Model Scale (CHBMS), developed by Champion in 1984 and revised in 1993, is used to measure women's beliefs about breast cancer and breast self-examination (BSE). The Turkish Version of the Champion's Health Belief Model Scale was validated by Gözüm and Aydın in 2004 with 8 sub-dimensions and 58 items. Questions were answered on a 5-point Likert-type response scale ranging from 1 (strongly disagree) to 5 (strongly agree), and mean scores were computed for each subscale. The total score that can be obtained from the scale is 58 minimum and 290 maximum. Thus, higher scores represent perceptions of greater susceptibility to breast cancer, greater benefits from screening, and higher barriers to screening. The opposite was expected for higher perceived barriers. A total scale score was also derived by computing the mean of the mean subscale scores, with barriers reverse coded.
The Health Belief Model Scale for Cervical Cancer and the Pap Smear Test(HBMSCCPS) | 4 Months
  Developed by Champion for breast cancer and mammography, this scale, which was adapted to cervical cancer and pap smear test by Güvenç, Akyüz, and Açıkel in 2011, is used to investigate the beliefs of women in respect of cervical cancer and the Pap Smear Test to assist healthcare professionals to develop more effective cervical cancer screening programmes. The scale consists of 35 items and five main dimensions. Questions were answered on a 5-point Likert-type response scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score that can be obtained from the scale is 35 minimum and 175 maximum. The higher scores indicate agreement with the beliefs of health assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah KÖK, Asst. Prof., Study Director — Department of Obstetrics and Gynecology Nursing, Gulhane Nursing Faculty, Health Sciences University

IPD SHARING:
Plan to Share IPD: No